CLINICAL TRIAL: NCT04941014
Title: Effects of Physical Activity on Quality of Life Among Female Undergraduate Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Health Education Research Foundation (HERF) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HERF/REC/2021-2
Record Dates: First submitted 2021-06-08; First posted 2021-06-28 (Actual); Last update posted 2021-06-28 (Actual); Status verified 2021-06

CONDITIONS: Quality of Life

STUDY DESIGN:
Intervention Model Description: Assignment
Who Masked: Participant
Masking Description: single
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Light Physical Activity (LPA) (Active Comparator): The guidelines from Rapid Assessment of Physical Activity (RAPA) participants were asked to perform Leisure Walk for 35 minutes
  Interventions: Behavioral: Light Physical Activity
- Moderate Physical Activity (MPA) (Active Comparator): The guidelines from Rapid Assessment of Physical Activity (RAPA) participants were asked to perform Brisk Walk for 30 minutes
  Interventions: Behavioral: Moderate Physical Activity
- Vigorous Physical activity (VPA) (Active Comparator): The guidelines from Rapid Assessment of Physical Activity (RAPA) participants were asked to perform jogging for 15 minutes
  Interventions: Behavioral: Vigourous Physical Activity

INTERVENTIONS:
Behavioral: Light Physical Activity — The guidelines from Rapid Assessment of Physical Activity (RAPA) participants were asked to perform Leisure Walk for 35 minutes
  Arms: Light Physical Activity (LPA)
Behavioral: Moderate Physical Activity — The guidelines from Rapid Assessment of Physical Activity (RAPA) participants were asked to perform Brisk Walk for 30 minutes
  Arms: Moderate Physical Activity (MPA)
Behavioral: Vigourous Physical Activity — The guidelines from Rapid Assessment of Physical Activity (RAPA) participants were asked to perform jogging for 15 minutes
  Arms: Vigorous Physical activity (VPA)

SUMMARY:
The main objective of the study is to determine the effects of physical activity on quality of life among female undergraduate students

ELIGIBILITY:
Inclusion Criteria:

-moderate level of academic stress measured on academic stress scale

Exclusion Criteria:

* students with diagnosed psychological disorders
* systematic diseases

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 52 (Actual)
Dates: Start 2019-05-04 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Quality of Life (QOL), | A change from baseline to six weeks of intervention will be observed
  The short form (SF-36) was used to observe Quality of Life (QOL), Minimum score is 0 and maximum is 100. maximum score indicate high quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Bilquis Postgraduate College for Women Pakistan Air force (PAF), Rawalpindi, Pakistan